CLINICAL TRIAL: NCT01031875
Title: Phase 2 Study With the Multi-Targeted Tyrosine-Kinase Inhibitor Pazopanib (GW786034) for Patients With Relapsed or Refractory Urothelial Cancer
Brief Title: Pazopanib Hydrochloride in Treating Patients With Metastatic Urethral Cancer or Bladder Cancer That Has Relapsed or Not Responded to Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ITA-MIL-IRCCS-INT-70/09; CDR0000661071 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2009-017093-20; EU-20990
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2012-09

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; stage IV bladder cancer; recurrent urethral cancer; distal urethral cancer; proximal urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; stage IV urethral cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Fluorodeoxyglucose F18

INTERVENTIONS:
Drug: pazopanib hydrochloride
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well pazopanib hydrochloride works in treating patients with or metastatic urothelial cancer or bladder cancer that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the activity of daily oral doses of pazopanib hydrochloride monotherapy in patients with relapsed/refractory metastatic urothelial carcinoma or transitional cell tumors.

Secondary

* To evaluate the safety and tolerability of pazopanib hydrochloride monotherapy in a population of chemotherapy pretreated patients.
* To assess progression-free survival of these patients.

Tertiary

* To evaluate the ability of whole-body 18FDG-PET to image metastases and monitor tumor response and to determine the rate of concordance with CT imaging and RECIST response criteria.
* To evaluate the relationship existing between tumor response measured by 18FDG-PET and progression-free survival.

OUTLINE: This is a multicenter study.

Patients receive oral pazopanib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo whole-body 18FDG-PET at baseline and periodically.

After completion of study treatment, patients are followed for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of transitional cell tumors of the bladder or the urothelium

  * Metastatic disease
  * Relapsed or refractory disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 2 cm by conventional techniques or ≥ 1 cm by spiral CT scan
* Must have failed ≥ 1 cisplatin-based conventional chemotherapy regimen for metastatic disease (neoadjuvant/adjuvant therapy excluded)
* No history or clinical evidence of CNS metastases or leptomeningeal carcinomatosis, except for individuals who were previously treated for CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for the past 6 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement)
* Alkaline phosphatase ≤ 4 x ULN
* Serum creatinine ≤ 1.5 mg/dL
* PT-INR/PTT < 1.5 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study therapy
* Able to swallow oral medication
* None of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Symptomatic peripheral vascular disease
  * NYHA class III or IV congestive heart failure
  * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted)
  * Uncontrolled hypertension
* No history of HIV infection or active chronic hepatitis B or C
* No active clinically serious infections > grade 2 NCI-CTC version 4.0
* No seizure disorder requiring medication (e.g., steroids or anti-epileptics)
* No history of any of the following conditions within the past 6 months:

  * Cerebrovascular accident
  * Pulmonary embolism
  * Untreated deep venous thrombosis
* No evidence or history of bleeding diathesis
* No known endobronchial lesions or involvement of large pulmonary vessels by tumor
* No hemoptysis within the past 6 weeks
* No gastrointestinal abnormalities that may increase the risk of GI bleeding or affect the absorption of investigational study drug
* No other cancer that is distinct in primary site or histology from the cancer being evaluated in this study, except cervical carcinoma in situ, treated basal cell carcinoma, or any cancer curatively treated > 5 years prior to study entry
* No substance abuse, medical, psychological, or social conditions that may interfere with the study participation or evaluation of the study results
* No concurrent unstable condition that could jeopardize patient safety and their compliance in the study
* No non-healing wound, fracture, or ulcer within the past 28 days
* No major trauma within the past 28 days
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib hydrochloride

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* At least 14 days since prior radiotherapy, except palliative radiotherapy
* At least 14 days since tumor embolization
* At least 14 days or 5 half-lives (whichever is longer) of a drug since prior chemotherapy, immunotherapy, biologic therapy, investigational therapy, or hormonal therapy
* At least 3 weeks since prior biologic response modifiers (e.g., G-CSF)

  * G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity (e.g., febrile neutropenia) when clinically indicated or at the discretion of the investigator, however they may not be used to avoid a required dose reduction
  * Chronic erythropoietin allowed provided no dose adjustment is undertaken within 2 months prior to the study or during the study
* No prior pazopanib hydrochloride
* No coronary artery by-pass graft surgery within the past 6 months
* No major surgery within the past 28 days
* Concurrent coumadin or heparin for therapeutic anticoagulation allowed provided that no prior evidence of underlying abnormality in PT-INR/PTT parameters exist
* Not concurrently undergoing renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial response) according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Safety and tolerability, in terms of incidence, nature, and severity of treatment-related adverse events according to CTCAE v4.0
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Salvioni, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Nicola Nicolai, MD — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Andrea Necchi, MD — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Result] Necchi A, Mariani L, Zaffaroni N, Schwartz LH, Giannatempo P, Crippa F, Morosi C, Lanocita R, Sava T, Ortega C, Messina C, Sacco C, Pennati M, Daidone MG, Nicolai N, De Braud F, Gianni AM, Salvioni R. Pazopanib in advanced and platinum-resistant urothelial cancer: an open-label, single group, phase 2 trial. Lancet Oncol. 2012 Aug;13(8):810-6. doi: 10.1016/S1470-2045(12)70294-2. Epub 2012 Jul 20. PMID 22819172